CLINICAL TRIAL: NCT01832597
Title: A Retrospective Multicenter Trial on Efficacy and Toxicity of Bendamustine Alone or Associated With Rituximab, As Salvage Therapy in Patients With Chronic Lymphoproliferative Disorders
Brief Title: Efficacy and Safety Study of Bendamustine With or Without Rituximab in Chronic Lymphoproliferative Disorders
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Studio Linfomi (Other)
Responsible Party: Sponsor
Other Study IDs: RetroBENDA
Record Dates: First submitted 2013-04-08; First posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Lymphocytic Leukaemia
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is collect and evaluate the clinical experience reached in Italy on the use of bendamustine alone or combined with rituximab as treatment of patients with relapsed or refractory chronic lymphoproliferative disorders.

DETAILED DESCRIPTION:
All patients who meet the criteria for inclusion will be included in the study. A specific database will be created to collect the following information: personal data, medical history, histology related to the underlying disease, comorbidities, laboratory data, initial staging, data on the dosage and the number of cycles administered, the recorded toxicity data, the clinical response and the main events (relapse, progression, death, and cause of death). These data will then be retrospectively examined in order to obtain information about the life-saving treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients with relapsed or refractory chronic lymphoproliferative disorders
* salvage treatment with Bendamustine +/- Rituximab
* age ≥ 18 years

Exclusion Criteria:

* previous treatment with Bendamustine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with relapsed or refractory chronic lymphoproliferative disorders treated with Bendamustine +/- Rituximab
Sampling Method: Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | At least 2 months after completion of therapy
  Evaluate the activity of Bendamustine +/- Rituximab in term of ORR

SECONDARY OUTCOMES:
Progression Free Survival (PFS) and Overall Survival (OS) | From the date of frist treatment cycle until the date of first documented progression or date of death for any cause, whichever came first, assessed up to 150 months
  Evaluate the activity of Bendamustine +/- Rituximab in term of PFS and OS
Number of Adverse Events | From the date of first tratment cycle until 6 months after the date of last treatment cycle
  Assess to efficacy of Bendamustine +/- Rituximab in term of grade III and IV National Cancer Institute Common Toxicity Criteria (NCI CTC) adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Luminari, MD, Study Director — Gruppi Italiano Studi Linfomi; Emilio Iannitto, MD, Principal Investigator — Gruppo Italiano Studio Linfomi
Locations (3):
- Italy (3):
  - UO di Ematologia, S.O. Annunziata, Cosenza, CZ
  - Dipartimento di Oncologia, Ematologia e Patologie dell'Apparato Respiratorio, Universita' di Modena e Reggio Emilia, Modena, MO
  - UO di Ematologia, AOUP Paolo Giaccone,, Palermo, PA

REFERENCES:
- [Background] Anderson JR, Cain KC, Gelber RD. Analysis of survival by tumor response. J Clin Oncol. 1983 Nov;1(11):710-9. doi: 10.1200/JCO.1983.1.11.710. PMID 6668489
- [Background] Anderson JR, Cain KC, Gelber RD. Analysis of survival by tumor response and other comparisons of time-to-event by outcome variables. J Clin Oncol. 2008 Aug 20;26(24):3913-5. doi: 10.1200/JCO.2008.16.1000. No abstract available. PMID 18711176
- [Background] Bergmann MA, Goebeler ME, Herold M, Emmerich B, Wilhelm M, Ruelfs C, Boening L, Hallek MJ; German CLL Study Group. Efficacy of bendamustine in patients with relapsed or refractory chronic lymphocytic leukemia: results of a phase I/II study of the German CLL Study Group. Haematologica. 2005 Oct;90(10):1357-64. PMID 16219572
- [Background] Cheson BD, Rummel MJ. Bendamustine: rebirth of an old drug. J Clin Oncol. 2009 Mar 20;27(9):1492-501. doi: 10.1200/JCO.2008.18.7252. Epub 2009 Feb 17. PMID 19224851
- [Background] Cheson BD, Wendtner CM, Pieper A, Dreyling M, Friedberg J, Hoelzer D, Moreau P, Gribben J, Knop S, Montillo M, Rummel M. Optimal use of bendamustine in chronic lymphocytic leukemia, non-Hodgkin lymphomas, and multiple myeloma: treatment recommendations from an international consensus panel. Clin Lymphoma Myeloma Leuk. 2010 Feb;10(1):21-7. doi: 10.3816/CLML.2010.n.002. PMID 20223726
- [Background] Ferrajoli A, Lee BN, Schlette EJ, O'Brien SM, Gao H, Wen S, Wierda WG, Estrov Z, Faderl S, Cohen EN, Li C, Reuben JM, Keating MJ. Lenalidomide induces complete and partial remissions in patients with relapsed and refractory chronic lymphocytic leukemia. Blood. 2008 Jun 1;111(11):5291-7. doi: 10.1182/blood-2007-12-130120. Epub 2008 Mar 11. PMID 18334676
- [Background] Oskolkova OV, Afonyushkin T, Leitner A, von Schlieffen E, Gargalovic PS, Lusis AJ, Binder BR, Bochkov VN. ATF4-dependent transcription is a key mechanism in VEGF up-regulation by oxidized phospholipids: critical role of oxidized sn-2 residues in activation of unfolded protein response. Blood. 2008 Jul 15;112(2):330-9. doi: 10.1182/blood-2007-09-112870. Epub 2008 May 1. PMID 18451308
- [Background] Foon KA, Hallek MJ. Changing paradigms in the treatment of chronic lymphocytic leukemia. Leukemia. 2010 Mar;24(3):500-11. doi: 10.1038/leu.2009.266. Epub 2009 Dec 24. PMID 20033051
- [Background] Forconi F, Fabbri A, Lenoci M, Sozzi E, Gozzetti A, Tassi M, Raspadori D, Lauria F. Low-dose oral fludarabine plus cyclophosphamide in elderly patients with untreated and relapsed or refractory chronic lymphocytic Leukaemia. Hematol Oncol. 2008 Dec;26(4):247-51. doi: 10.1002/hon.868. PMID 18642397
- [Background] Giannopoulos K, Dmoszynska A, Kowal M, Wasik-Szczepanek E, Bojarska-Junak A, Rolinski J, Dohner H, Stilgenbauer S, Bullinger L. Thalidomide exerts distinct molecular antileukemic effects and combined thalidomide/fludarabine therapy is clinically effective in high-risk chronic lymphocytic leukemia. Leukemia. 2009 Oct;23(10):1771-8. doi: 10.1038/leu.2009.98. Epub 2009 May 14. PMID 19440214
- [Background] Gribben JG. How I treat CLL up front. Blood. 2010 Jan 14;115(2):187-97. doi: 10.1182/blood-2009-08-207126. Epub 2009 Oct 22. PMID 19850738
- [Background] Hallek M, Schmitt B, Wilhelm M, Busch R, Krober A, Fostitsch HP, Sezer O, Herold M, Knauf W, Wendtner CM, Kuse R, Freund M, Franke A, Schriever F, Nerl C, Dohner H, Thiel E, Hiddemann W, Brittinger G, Emmerich B; German Chronic Lymphocytic Leukaemia Study Group. Fludarabine plus cyclophosphamide is an efficient treatment for advanced chronic lymphocytic leukaemia (CLL): results of a phase II study of the German CLL Study Group. Br J Haematol. 2001 Aug;114(2):342-8. doi: 10.1046/j.1365-2141.2001.02959.x. PMID 11529853
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Background] Knauf WU, Lissichkov T, Aldaoud A, Liberati A, Loscertales J, Herbrecht R, Juliusson G, Postner G, Gercheva L, Goranov S, Becker M, Fricke HJ, Huguet F, Del Giudice I, Klein P, Tremmel L, Merkle K, Montillo M. Phase III randomized study of bendamustine compared with chlorambucil in previously untreated patients with chronic lymphocytic leukemia. J Clin Oncol. 2009 Sep 10;27(26):4378-84. doi: 10.1200/JCO.2008.20.8389. Epub 2009 Aug 3. PMID 19652068
- [Background] Lamanna N, Kalaycio M, Maslak P, Jurcic JG, Heaney M, Brentjens R, Zelenetz AD, Horgan D, Gencarelli A, Panageas KS, Scheinberg DA, Weiss MA. Pentostatin, cyclophosphamide, and rituximab is an active, well-tolerated regimen for patients with previously treated chronic lymphocytic leukemia. J Clin Oncol. 2006 Apr 1;24(10):1575-81. doi: 10.1200/JCO.2005.04.3836. Epub 2006 Mar 6. PMID 16520464
- [Background] Leoni LM, Bailey B, Reifert J, Bendall HH, Zeller RW, Corbeil J, Elliott G, Niemeyer CC. Bendamustine (Treanda) displays a distinct pattern of cytotoxicity and unique mechanistic features compared with other alkylating agents. Clin Cancer Res. 2008 Jan 1;14(1):309-17. doi: 10.1158/1078-0432.CCR-07-1061. PMID 18172283
- [Background] Lin TS, Ruppert AS, Johnson AJ, Fischer B, Heerema NA, Andritsos LA, Blum KA, Flynn JM, Jones JA, Hu W, Moran ME, Mitchell SM, Smith LL, Wagner AJ, Raymond CA, Schaaf LJ, Phelps MA, Villalona-Calero MA, Grever MR, Byrd JC. Phase II study of flavopiridol in relapsed chronic lymphocytic leukemia demonstrating high response rates in genetically high-risk disease. J Clin Oncol. 2009 Dec 10;27(35):6012-8. doi: 10.1200/JCO.2009.22.6944. Epub 2009 Oct 13. PMID 19826119
- [Background] Lissitchkov T, Arnaudov G, Peytchev D, Merkle Kh. Phase-I/II study to evaluate dose limiting toxicity, maximum tolerated dose, and tolerability of bendamustine HCl in pre-treated patients with B-chronic lymphocytic leukaemia (Binet stages B and C) requiring therapy. J Cancer Res Clin Oncol. 2006 Feb;132(2):99-104. doi: 10.1007/s00432-005-0050-z. Epub 2005 Nov 15. PMID 16292542
- [Background] Mossner E, Brunker P, Moser S, Puntener U, Schmidt C, Herter S, Grau R, Gerdes C, Nopora A, van Puijenbroek E, Ferrara C, Sondermann P, Jager C, Strein P, Fertig G, Friess T, Schull C, Bauer S, Dal Porto J, Del Nagro C, Dabbagh K, Dyer MJ, Poppema S, Klein C, Umana P. Increasing the efficacy of CD20 antibody therapy through the engineering of a new type II anti-CD20 antibody with enhanced direct and immune effector cell-mediated B-cell cytotoxicity. Blood. 2010 Jun 3;115(22):4393-402. doi: 10.1182/blood-2009-06-225979. Epub 2010 Mar 1. PMID 20194898
- [Background] Motta M, Wierda WG, Ferrajoli A. Chronic lymphocytic leukemia: treatment options for patients with refractory disease. Cancer. 2009 Sep 1;115(17):3830-41. doi: 10.1002/cncr.24479. PMID 19536902
- [Background] O'Brien SM, Kantarjian HM, Cortes J, Beran M, Koller CA, Giles FJ, Lerner S, Keating M. Results of the fludarabine and cyclophosphamide combination regimen in chronic lymphocytic leukemia. J Clin Oncol. 2001 Mar 1;19(5):1414-20. doi: 10.1200/JCO.2001.19.5.1414. PMID 11230486
- [Background] Robak T, Dmoszynska A, Solal-Celigny P, Warzocha K, Loscertales J, Catalano J, Afanasiev BV, Larratt L, Geisler CH, Montillo M, Zyuzgin I, Ganly PS, Dartigeas C, Rosta A, Maurer J, Mendila M, Saville MW, Valente N, Wenger MK, Moiseev SI. Rituximab plus fludarabine and cyclophosphamide prolongs progression-free survival compared with fludarabine and cyclophosphamide alone in previously treated chronic lymphocytic leukemia. J Clin Oncol. 2010 Apr 1;28(10):1756-65. doi: 10.1200/JCO.2009.26.4556. Epub 2010 Mar 1. PMID 20194844
- [Background] Tageja N, Nagi J. Bendamustine: something old, something new. Cancer Chemother Pharmacol. 2010 Aug;66(3):413-23. doi: 10.1007/s00280-010-1317-x. Epub 2010 Apr 8. PMID 20376452
- [Background] Wierda W, O'Brien S, Wen S, Faderl S, Garcia-Manero G, Thomas D, Do KA, Cortes J, Koller C, Beran M, Ferrajoli A, Giles F, Lerner S, Albitar M, Kantarjian H, Keating M. Chemoimmunotherapy with fludarabine, cyclophosphamide, and rituximab for relapsed and refractory chronic lymphocytic leukemia. J Clin Oncol. 2005 Jun 20;23(18):4070-8. doi: 10.1200/JCO.2005.12.516. Epub 2005 Mar 14. PMID 15767647
- [Background] Wierda WG, Kipps TJ, Mayer J, Stilgenbauer S, Williams CD, Hellmann A, Robak T, Furman RR, Hillmen P, Trneny M, Dyer MJ, Padmanabhan S, Piotrowska M, Kozak T, Chan G, Davis R, Losic N, Wilms J, Russell CA, Osterborg A; Hx-CD20-406 Study Investigators. Ofatumumab as single-agent CD20 immunotherapy in fludarabine-refractory chronic lymphocytic leukemia. J Clin Oncol. 2010 Apr 1;28(10):1749-55. doi: 10.1200/JCO.2009.25.3187. Epub 2010 Mar 1. PMID 20194866
- [Background] Zenz T, Mertens D, Kuppers R, Dohner H, Stilgenbauer S. From pathogenesis to treatment of chronic lymphocytic leukaemia. Nat Rev Cancer. 2010 Jan;10(1):37-50. doi: 10.1038/nrc2764. Epub 2009 Dec 3. PMID 19956173